CLINICAL TRIAL: NCT03170869
Title: SPEED 1 Trial: Bridge to Orthotopic Liver Transplantation (OLT) - (Surefire Precision vs Endhole Embolization With DEBTACE)
Brief Title: Bridge to Orthotopic Liver Transplantation (OLT) - Surefire Precision vs Endhole Embolization With DEBTACE
Acronym: SPEED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor withdrew funding
Sponsor: University of Colorado, Denver (Other)
Collaborators: Surefire Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-1313.cc
Record Dates: First submitted 2017-05-26; First posted 2017-05-31 (Actual); Results first posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Hepatocellular Carcinoma of the Liver; Subjects Eligible for Liver Transplantation

STUDY DESIGN:
Intervention Model Description: Fifty (50) subjects will be enrolled in the prospective arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- DEB-TACE Procedure with Surefire Precision Infusion System (Experimental): The study duration for each patient is 24 months and includes a baseline visit, procedure visit and follow-up visits at 1 week, 1 month, 3 months, 6 months and every 3 months until liver transplant or death.
  The following evaluations/activities will be performed at baseline: Informed consent, history, physical exam, data collection of CT/ MRI within 1 month of the visit date, data collection of lab values and quality of life questionnaire.
  The treatment visit includes the DEB-TACE procedure with the Surefire Precision Infusion System. After the procedure, a Cone Beam CT of the liver will be performed to determine distribution and density of the beads in the tumor and adverse events monitoring.
  The following evaluations / activities will be performed during the follow-up period: physical exam, data collection of contrast enhanced CT/MRI to evaluate tumor response, data collection of lab values, adverse event monitoring and quality of life questionnaire.
  Interventions: Device: Surefire Precision Infusion System

INTERVENTIONS:
Device: Surefire Precision Infusion System — All patients enrolled in this protocol will receive DEB-TACE, which is the standard of care prescribed by their physician. Standard 5 Fr and 3 Fr catheters will be used to perform diagnostic angiography to map the hepatic vasculature to the tumor. Using standard technique, the target vessel feeding the tumor will be catheterized and DEB-TACE administered using the Surefire Precision catheter. The Doxorubicin dosing used in the DEB-TACE will be based upon tumor volume. DEB-TACE will be administered until the first of the following endpoints are reached: Achievement of target dose with stasis, leeching of contrast through the expandable tip and development of distal intrahepatic collaterals.

SUMMARY:
The purpose of this study will be to prospectively evaluate the outcomes of patients with hepatocellular carcinoma (HCC) who undergo DEB-TACE (drug-eluting bead trans-arterial chemoembolization) with the Surefire Precision Infusion System for intentional effect of down-staging patients to OLT.

Patients with HCC and who are considered candidates for liver transplantation but outside Milancriteria and meet the eligibility criteria will be enrolled in the prospective single arm study.

Results of the prospective cohort will be compared to matched historical control patients who were previously treated with DEB-TACE, delivered with standard endhole catheters. This includes all patients treated at the University of Colorado since 2009 treated with 100-300 micron beads for whom follow-up is available.

DETAILED DESCRIPTION:
This is a single institution prospective clinical trial with historical matched controls. This protocol standardizes DEB-TACE delivery with the Surefire Precision Infusion System. This protocol does not change patient therapy. All patient safety monitoring, treatment procedures and follow-up procedures will be performed in accordance with standard clinical practice.

Fifty (50) subjects will be enrolled in the prospective arm. Data from one hundred (100) historical randomly sampled control subjects (1:2 ratio) will be selected.

Subjects will be followed at 1 week, 1 month, 3 months, then every 3 months, following the initial DEB-TACE procedure until the subject receives a liver transplant or death. The study will be concluded upon completion of enrollment and follow-up of the 50 patients. It is estimated that the time to complete patient enrollment and follow-up is 24 months. The estimated date for study completion (complete primary analyses) is June 2018. This is based on the average survival vs. time to transplant at this center. If there are individual patients that extend beyond this period the time may be slightly extended.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older with the diagnosis of HCC currently being evaluated for liver transplantation and considered for downstaging.
* Patients undergoing Surefire DEB-TACE procedure as clinically determined
* Single tumor that is >5 cm and less than 8 cm, OR 1 to 3 tumors with combined diameter greater than 15 cm and less than 24 cm
* No portal invasion or extrahepatic spread
* No previous chemotherapy, radiotherapy or transarterial embolization (with or without chemotherapy)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Preserved liver function (Child-Pugh Class A or B).
* Discrete hepatic artery feeding the tumor with vessel diameter > 1.5 mm

Exclusion Criteria:

* Advanced bilirubin levels > 3 mg/dl
* AST or ALT>5 upper limit of normal or >250 U/l
* Advanced tumoral disease, defined as vascular invasion, extrahepatic spread, or diffuse HCC (50% liver involvement)
* Contraindications for doxorubicin administration.
* Child's Class C
* Vessels providing flow to the tumor that are less than 1.5 mm in diameter

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2018-09-11 (Actual); Study Completion 2018-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David T Johnson, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DEB-TACE Procedure With Surefire Precision Infusion System
Started | 11
Completed | 3
Not Completed | 8
Not completed — Protocol Violation | 5
Not completed — Early study termination | 3

BASELINE CHARACTERISTICS:
Arm/Group | DEB-TACE Procedure With Surefire Precision Infusion System
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 60.27 [42 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Local Recurrence Rate (LRR)
Description: For the outcome of local recurrence rate (LRR) we will test the null hypothesis of no difference in the proportion of patients with local recurrence by catheter type using a Fisher's exact test.
Time Frame: 6 months
Population: Zero participants analyzed as the study was terminated prior to data for outcome measures to be assessed. No data was collected or analyzed for this outcome measure.
Groups:
- DEB-TACE Procedure With Surefire Precision Infusion System: The study duration for each patient is 24 months and includes a baseline visit, procedure visit and follow-up visits at 1 week, 1 month, 3 months, 6 months and every 3 months until liver transplant or death.
  The following evaluations/activities will be performed at baseline: Informed consent, history, physical exam, data collection of CT/ MRI within 1 month of the visit date, data collection of lab values and quality of life questionnaire.
  The treatment visit includes the DEB-TACE procedure with the Surefire Precision Infusion System. After the procedure, a Cone Beam CT of the liver will be performed.
  The following evaluations / activities will be performed during the follow-up period: physical exam, data collection of contrast enhanced CT/MRI to evaluate tumor response, data collection of lab values, adverse event monitoring and quality of life questionnaire.
Arm/Group | DEB-TACE Procedure With Surefire Precision Infusion System
Number analyzed (Participants) | 0

2. Secondary Outcome: Tumor Response
Description: For the outcome of tumor response measured as the change in enhancing tumor size (pretreatment - post treatment) we will evaluate changes at 1 month and 6 month separately.
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | DEB-TACE Procedure With Surefire Precision Infusion System
Number analyzed (Participants) | 0

3. Secondary Outcome: Time to Progression
Description: For the outcome of time to progression, we will quantify the number of weeks from treatment until tumor progression.
Time Frame: Every 3 months through 24 months
Population: Zero participants analyzed as the study was terminated. No data was collected or analyzed for this outcome measure.
Arm/Group | DEB-TACE Procedure With Surefire Precision Infusion System
Number analyzed (Participants) | 0

4. Secondary Outcome: Survival Time
Description: For the outcome of survival time, we will quantify the number of weeks from treatment until death.
Time Frame: Every 3 months through 24 months
Population: as for outcome 1
Arm/Group | DEB-TACE Procedure With Surefire Precision Infusion System
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months from the baseline procedure with the Surefire device
Arm/Group | DEB-TACE Procedure With Surefire Precision Infusion System
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 2/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DEB-TACE Procedure With Surefire Precision Infusion System (N=11)
Abdominal pain (Hepatobiliary disorders) | 1
Infection (General disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DEB-TACE Procedure With Surefire Precision Infusion System (N=11)
Flow limiting dissection of the anterior right hepatic artery (Hepatobiliary disorders) | 1
Abdominal pain (General disorders) | 6
Nausea (General disorders) | 5
Fatigue (General disorders) | 5
Chest pain during sleep (General disorders) | 1
Elevated AFP levels (General disorders) | 2
Occasional hot flashes (General disorders) | 2
Mild groin paint post re-treatment (General disorders) | 2
Elevated Hep C Quantitative PCR (General disorders) | 1
Muscle wasting (General disorders) | 2
Abdominal distention (General disorders) | 3
Edema (General disorders) | 3
Admission for infection (General disorders) | 2
Increased AFib (General disorders) | 1
Blood bilirubin increased (General disorders) | 2
Hypoalbuminemia (General disorders) | 2
Elevated INR levels (General disorders) | 2
Headaches (General disorders) | 1
Fever and chills (General disorders) | 2
Post embolization sydrome (General disorders) | 2
Difficulty with pain control (General disorders) | 1
Elevated AFP levels (General disorders) | 1
Elevated lactate whole blood venous levels (General disorders) | 3
Cough and chest tightness (General disorders) | 1
Platelet count decreased (General disorders) | 1
Encephalopathy (General disorders) | 2
Elevated ammonia levels (General disorders) | 1
Dizziness (General disorders) | 1
Acute kidney injury (General disorders) | 1
Hyperkalemia (General disorders) | 1
Constipation (General disorders) | 1
Depression (General disorders) | 1
Ascites (General disorders) | 1

LIMITATIONS AND CAVEATS:
Zero participants were analyzed as the study was terminated early due to change in funding. No statistical analysis was performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/69/NCT03170869/Prot_SAP_000.pdf